CLINICAL TRIAL: NCT03191994
Title: Exercise Promotes Neuroplasticity in Depressed and Healthy Brains: An fMRI Pilot Study
Brief Title: Impact of an Eight Week Exercise Intervention in Treating Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ontario Institute of Technology (Other)
Responsible Party: Principal Investigator, Bernadette Murphy, Professor, University of Ontario Institute of Technology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UOntarioIT
Record Dates: First submitted 2017-06-08; First posted 2017-06-19 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: MDD exercise group, MDD control group, Healthy exercise group, Healthy control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MDD exercise group (Experimental): This group will receive eight weeks of moderate exercise in addition to their usual treatment
  Interventions: Behavioral: Exercise
- MDD control group (No Intervention): This group will receive usual care with no exercise
- Healthy Exercise (Experimental): This group will perform an eight week moderate intensity exercise intervention
  Interventions: Behavioral: Exercise
- Healthy control (No Intervention): This group will not perform exercise

INTERVENTIONS:
Behavioral: Exercise — a structured, supervised eight week moderate intensity exercise intervention
  Arms: Healthy Exercise; MDD exercise group

SUMMARY:
To investigate the impact of a structured eight week exercise intervention as an add-on therapy in treating Major Depressive Disorder. Using behavioural techniques and neuroimaging to measure changes in brain function following an exercise intervention in people with clinical depression. By correlating changes in the hippocampus with changes in HPA axis hormones, inflammatory cytokines and growth factors it is possible to determine which of the biochemical markers is most predictive of improved neural function.

DETAILED DESCRIPTION:
Memory impairment is the most frequently reported cognitive symptom in people with depression. However, research in this area has presented mixed findings in terms of the type, severity and specificity of memory deficits. One finding that has been well established is the impairment in episodic memory (memory for a specific past experience in one's life) with a sparing of semantic memory (present knowledge of universal truths such as "the sky is blue"), and short-term memory. Behavioural and neuroimaging studies investigating the stage of the memory deficit in people with depression have found that both the encoding and retrieval processes are impaired. Although the neural underpinnings of impaired memory in MDD are not completely understood, the majority of evidence implicates abnormal activity in the hippocampal region critical for normal memory formation.

Exercise for depression has been a common research theme for the past several years however its mechanism of action remains unknown. Many studies have reported higher levels of cardiorespiratory fitness and increased habitual physical activity being associated with lower depressive symptomatology and greater emotional well-being, while lower levels of cardiorespiratory fitness being associated with increased risk of developing depressive illness. Exercise alone or in combination with other treatment options, such as pharmacotherapy or cognitive behavioural therapy have all been effective in treating depression with response rates for exercise being comparable to these mainstream therapies. Exercise protects against the development of neurodegenerative diseases delays the negative effects of aging and improves sleep quality. Exercise also reduces inflammation, normalizes cortisol secretion, increases hippocampal neurogenesis, increases cerebrovascular perfusion, improves the structure and function of the hippocampus, facilitates neurocognitive recovery from traumatic brain injury reverses brain volume loss in elderly and schizophrenic individuals and improves learning and memory. These findings suggest that the relationship between fitness and cognition is partly mediated by processes that involve cerebral circulation. These positive effects of exercise on neuroanatomy and vascularization can be partly explained by the interactive cascade of growth factor signalling associated with exercise that increases the ability of cerebral blood vessels to respond to demand. Habitual exercise is an effective way to improve endothelial function by increasing arterial compliance and decreasing arterial stiffness, oxidative stress, and vascular inflammation.

The overall goal of this research study is to investigate the effects of a well-defined, structured, supervised exercise program on brain function in healthy and clinically depressed individuals. This research aims to fill the gaps in the literature by elucidating the anti-depressant mechanisms which exercise targets and if these effects parallel young healthy sedentary individuals.

To investigate the effects of a moderate-intensity structured, supervised 8 week exercise program in people with MDD when combined with a Mental Health Day Treatment (MHDT) program, as compared to the MHDT on its own. All outcome measures will be assessed at baseline and 8 weeks. A non-depressed exercise control group will be used to compare the effects of exercise in depressed and non-depressed individuals:

i. depressive symptoms ii. anxiety iii. sleep quality iv. plasma IL-1β, IL-1ra, IL-6, IFN-γ, TNF-α and IL-10, BDNF v. salivary cortisol vi. performance on an associative memory task and concomitant fMRI hippocampal activation.

ELIGIBILITY:
Inclusion Criteria:

* all participants must have no contraindications to exercise, be considered 'low active' (exercise less than 3 times per week for less than 20 minutes), MRI safe MDD group must be diagnosed by psychiatrist based on DSM-V criteria and pharmacological medication stabilized for a minimum of 6 weeks

Exclusion Criteria:

* no immune disorders

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-01-02; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Brain function during an associative memory task | eight weeks
  Participants will be MRI safety screened to ensure no metal implants. Using fMRI to determine brain activity during an associative memory task. Participants will be scanned on a 3-Tesla MR scanner. Scans will be acquired in the oblique coronal plane of the hippocampus. 416 functional scans will be acquired with a T2*-weighted gradient EPI sequence. Preprocessing will be performed using Statistical Parametric Mapping. General linear model will be performed at the single-subject level and statistical contrasts will be created modeling the hemodynamic response function of correct and incorrect responses. Random effects analysis will be performed using the contrast of t-test of correct > incorrect. Significant clusters from an independent samples t-test for correct>incorrect at baseline will be used to extract contrast beta values for correct>incorrect in pre and post scans. Average beta values will be imported into SPSS and a 2 x 2 repeated measures ANOVA (group x time).

SECONDARY OUTCOMES:
Depression scores | eight weeks
  Depression severity was determined using the self-reported Beck Depression Inventory (BDI). The BDI measures depression severity ranging from mile to severe depression. The higher the score the greater the depression severity.
Biochemical markers | eight weeks
  Peripheral venous blood will be collected from each participant at baseline and eight weeks by venipuncture into ethylenediaminetetraacetic acid (EDTA) tubes. Plasma proteins IL-1β, IL-1Ra, IL-6, IL-10 TNF-α, BDNF and total CTHB will be quantified using enzyme-linked immunosorbant assays (ELISA) following manufacturer's protocols (R&D Systems, MN, USA; BioLegend, CA, USA). Cortisol was measured using participant saliva and quantified using ELISA. Outcome measures will be measured in picograms/ml
Sleep quality | eight weeks
  Sleep quality will be measured using the Pittsburgh Sleep Quality Index a (PSQI) a self reported questionnaire. Sleep quality over the score over 5 is indicative of poor sleep quality.
Anxiety | eight weeks
  Anxiety will be measured using the Hospital Anxiety Depression Scale (HADS) a self-reported questionnaire. The higher the score the greater the anxiety severity.
Memory performance | eight weeks
  Associated memory task using face and names pairs. This was performed during the fMRI. Outcome measures include correct and incorrect reponses

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette Murphy, PhD, Principal Investigator — University of Ontario Institute of Technology
Locations (1):
- University of Ontario Institute of Technology, Oshawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Airaksinen E, Larsson M, Lundberg I, Forsell Y. Cognitive functions in depressive disorders: evidence from a population-based study. Psychol Med. 2004 Jan;34(1):83-91. doi: 10.1017/s0033291703008559. PMID 14971629
- [Background] Blumenthal JA, Babyak MA, Doraiswamy PM, Watkins L, Hoffman BM, Barbour KA, Herman S, Craighead WE, Brosse AL, Waugh R, Hinderliter A, Sherwood A. Exercise and pharmacotherapy in the treatment of major depressive disorder. Psychosom Med. 2007 Sep-Oct;69(7):587-96. doi: 10.1097/PSY.0b013e318148c19a. Epub 2007 Sep 10. PMID 17846259
- [Background] Blumenthal JA, Babyak MA, Moore KA, Craighead WE, Herman S, Khatri P, Waugh R, Napolitano MA, Forman LM, Appelbaum M, Doraiswamy PM, Krishnan KR. Effects of exercise training on older patients with major depression. Arch Intern Med. 1999 Oct 25;159(19):2349-56. doi: 10.1001/archinte.159.19.2349. PMID 10547175
- [Background] Cotman CW, Berchtold NC, Christie LA. Exercise builds brain health: key roles of growth factor cascades and inflammation. Trends Neurosci. 2007 Sep;30(9):464-72. doi: 10.1016/j.tins.2007.06.011. Epub 2007 Aug 31. PMID 17765329
- [Background] Davenport MH, Hogan DB, Eskes GA, Longman RS, Poulin MJ. Cerebrovascular reserve: the link between fitness and cognitive function? Exerc Sport Sci Rev. 2012 Jul;40(3):153-8. doi: 10.1097/JES.0b013e3182553430. PMID 22504726
- [Background] Erickson KI, Miller DL, Roecklein KA. The aging hippocampus: interactions between exercise, depression, and BDNF. Neuroscientist. 2012 Feb;18(1):82-97. doi: 10.1177/1073858410397054. Epub 2011 Apr 29. PMID 21531985
- [Background] Erickson KI, Voss MW, Prakash RS, Basak C, Szabo A, Chaddock L, Kim JS, Heo S, Alves H, White SM, Wojcicki TR, Mailey E, Vieira VJ, Martin SA, Pence BD, Woods JA, McAuley E, Kramer AF. Exercise training increases size of hippocampus and improves memory. Proc Natl Acad Sci U S A. 2011 Feb 15;108(7):3017-22. doi: 10.1073/pnas.1015950108. Epub 2011 Jan 31. PMID 21282661
- [Background] Pajonk FG, Wobrock T, Gruber O, Scherk H, Berner D, Kaizl I, Kierer A, Muller S, Oest M, Meyer T, Backens M, Schneider-Axmann T, Thornton AE, Honer WG, Falkai P. Hippocampal plasticity in response to exercise in schizophrenia. Arch Gen Psychiatry. 2010 Feb;67(2):133-43. doi: 10.1001/archgenpsychiatry.2009.193. PMID 20124113
- [Derived] Gourgouvelis J, Yielder P, Murphy B. Exercise Promotes Neuroplasticity in Both Healthy and Depressed Brains: An fMRI Pilot Study. Neural Plast. 2017;2017:8305287. doi: 10.1155/2017/8305287. Epub 2017 Jul 30. PMID 28828187